CLINICAL TRIAL: NCT03284866
Title: A Randomized, Placebo-Controlled Trial of HPV Vaccination to Reduce Cervical High-Grade Squamous Intraepithelial Lesions Among HIV-Infected Women Participating in an HPV Test-and-Treat Program (COVENANT)
Brief Title: HPV Vaccine Therapy in Reducing High-Grade Cervical Lesions in Patients With HIV and HPV
Acronym: COVENANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); University of Arkansas (Other); AIDS and Cancer Specimen Resource (Other); Merck Sharp & Dohme LLC (Industry); The Emmes Company, LLC (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AMC-099; NCI-2016-00841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-099 (Other: AIDS Malignancy Consortium); AMC-099 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-09-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: AIDS-Related Human Papillomavirus Infection; High Grade Cervical Squamous Intraepithelial Neoplasia; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I, recombinant HPV 9-valent vaccine (Experimental): Patients receive Recombinant Human Papillomavirus Nonavalent Vaccine (Gardasil 9) IM at baseline, 4, and 26 weeks in the absence of disease progression or unacceptable toxicity, with sample collection for Laboratory Biomarker Analysis.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm II, saline (Placebo Comparator): Patients receive saline placebo vaccine IM at baseline, 4, and 26 weeks, with sample collection for Laboratory Biomarker Analysis.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Saline

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine; Recombinant HPV 9-valent Vaccine
  Arms: Arm I, recombinant HPV 9-valent vaccine
Other: Saline — Given IM
  Other Names: Sodium Chloride 0.9%
  Arms: Arm II, saline

SUMMARY:
This randomized phase III trial studies how well human papillomavirus (HPV) vaccine therapy works in reducing high-grade cervical lesions in patients with human immunodeficiency virus (HIV) and HPV. Vaccines made from HPV peptides or antigens may help the body build an effective immune response to kill the HPV virus and prevent cervical lesions from developing or coming back after being removed.

DETAILED DESCRIPTION:
At screening, potential participants will be tested for cervical human papillomavirus (HPV) infection (GeneXpert hrHPV assay and HPV DNA PCR) and undergo cervical colposcopy to confirm the absence of cervical cancer. If eligible, the participant will be randomized to receive either the 9-valent HPV vaccine or saline placebo.

Participants will return 4 and 26 weeks later for the second dose of vaccine or placebo. At week 4, participants will have cervical colposcopy and undergo cryotherapy or loop electrosurgical excisional procedure (LEEP) as appropriate. Participants undergoing cervical cryotherapy will have cervical biopsies before the treatment. Participants will be followed with HPV testing (Gene Xpert and HPV DNA PCR) at weeks 26, 52, 78, and 104, and will have cervical cytology and colposcopy with biopsies at weeks 26, 52, and 104.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load, or documentation of receipt of antiretroviral therapy; Note: the term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally; WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment; a reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a western blot or a plasma HIV-1 RNA viral load
* HPV positive by the GeneXpert hrHPV assay with HPV16, HPV 18/45, or HPV31/33/35/52/58 detected; Note: participants who are hrHPV positive with only HPV51/59 or HPV 39/68/56/66 detected are not eligible
* Receipt of ART for at least 180 days prior to randomization
* Participants of childbearing potential, defined as a sexually mature woman who: (1) has not undergone a hysterectomy or bilateral oophorectomy or (2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must have a negative urine or serum pregnancy test within 3 weeks prior to enrollment and agree to use an effective form of contraception (e.g., barrier contraception or hormonal contraception), delaying pregnancy for at least 12 months and ideally for the duration of the study; Note: those willing to participate delay pregnancy for at least 6 months, while receiving the recombinant human papillomavirus nonavalent (9vHPV) vaccine (or placebo)
* If the participant is of childbearing potential, she should be at least 3 months postpartum
* Karnofsky score >= 70%
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current sexually transmitted infection (STI) requiring treatment (women may participate after adequate treatment, at the discretion of the treating provider)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Gardasil or Gardasil 9
* Uncontrolled intercurrent illness that would limit compliance with study requirements
* Prior hysterectomy with removal of the cervix
* Prior treatment for cervical HSIL
* Prior history of cervical, vulvar, or vaginal cancer
* Cervical, vulvar, or vaginal lesions suspicious for cancer based on clinical appearance (e.g. necrotic, ulcerated, and/or fungating masses), unless biopsies show no invasive cancer
* Known bleeding diathesis
* Prior HPV vaccination
* Current or planned use of anticoagulants other than aspirin or non-steroidal anti-inflammatory agents

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of cervical high-grade squamous intraepithelial lesions (HSIL) or cervical cancer | After week 4 study visit to week 52 post-randomization
  For each arm (vaccine and placebo), the event rate will be estimated using its point estimate and 95% Poisson confidence intervals. Poisson regression analyses will be used to compare the two arms with respect to event rate. In addition, time to event from week 4 to 52 will be described using the Kaplan-Meier method for each arm, and the two arms will be compared with respect to time to event using the log-rank test.

SECONDARY OUTCOMES:
Occurrence of cervical HSIL from weeks 52-104 | After week 52 to week 104
  The event rate for each arm from week 52 to week 104 for women who are event-free at 52 weeks will be estimated using its point estimate and 95% Poisson confidence interval. Poisson regression will be used to compare the two groups with respect to the event rate from week 52 to 104.
Role of baseline types and quantity of HPV as predictors of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if baseline HPV types are associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of presence of HSIL at baseline as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if the presence of HSIL at baseline is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of CD4+ cell count as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if baseline CD4+ cell count is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of plasma HIV-1 RNA as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if baseline plasma HIV-1 RNA count is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of ART use as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if ART use is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of age as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if age is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of sexual behavior as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if sexual behavior is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Role of vaccination use as a predictor of sustained absence | At baseline and week 4
  Poisson regression analyses will be used to determine if vaccine use is associated with of sustained absence of cervical HSIL and clearance of HPV infections after cryotherapy or LEEP. This analysis will also control for use of LEEP or cryotherapy.
Incident cervical vaccine type HPV infections defined as infections at 2 consecutive timepoints and assessed using type specific HPV DNA polymerase chain reaction (PCR) | Up to week 104
  Vaccine and placebo participants will be compared with respect to these proportions using the chi-square test corrected for continuity.
Abnormal cervical cytology | Baseline, week 26, 52, and 104
  The proportion of women with abnormal cervical cytology at baseline, week 26, 52, and 104 will be reported and compared between arms.
Prevalent vulvar HSIL or cancer | Up to week 4
  The prevalence of vulvar HSIL or cancer at baseline will be estimated using the binomial proportion and its 95% confidence interval.
Incident vulvar HSIL or cancer | Up to week 104
  The proportion of women who acquire vulvar HSIL or cancer among those negative for vulvar HSIL or cancer at baseline for both intervention arms will be estimated as a binomial proportion for both groups. The chi-square test corrected for continuity will be used to compare arms with respect to the proportions who acquire vulvar HSIL during the study.
Clinical and demographic factors associated with incident vulvar HSIL or cancer | Up to week 104
  Logistic regression analyses will be used to evaluate associations with incident vulvar HSIL or cancer acquisition with clinical and demographic factors and arm.

OTHER OUTCOMES:
HPV type distributions | Up to week 104
  Will characterize the HPV type distribution in baseline histology specimens and compare this to the types observed among incident cervical and vulvar HSIL lesions. Specifically, will compare the number and proportion of vaccine-type and non-vaccine type lesions between arms.
HPV strain variant analysis of cervical and vulvar HSIL specimens | Up to week 104
  For study participants who have the same HPV type in HSIL specimens at baseline and follow-up time points, sequencing will be performed to determine whether or not HSIL is caused by an identical HPV strain. Will use all available pairs of baseline and follow-up HSIL caused by the same HPV type. Will report the proportion of these pairs with the same HPV strain in both treatment arms. Additionally, will report the rates of HSIL caused by new vaccine type infections. We will compare the two study groups using a chi-square test. This will be a descriptive analysis only as no sufficient data on which to power this analysis.
Tissue microarray library of cervical specimens for biomarker analysis and discovery | Up to week 104
  Specimen banking objective. There is no pre-specified statistical analysis plan for this objective. Any future studies using these specimens will need to receive separate approval by NCI and CTEP.
hrHPV type distribution in the anus | Up to week 104
  McNemar's chi-square test to compare the prevalence of that type in the anus and cervix will be used. For each hrHPV type, chi-square analyses will be used to compare the two HPV vaccination groups with respect to the distribution of that type in the (anus, cervix). Will report the proportion of incident cervical infections that were preceded by anal detection of the same type.
hrHPV type prevalence in the anus | Up to week 104
  McNemar's chi-square test to compare the prevalence of that type in the anus and cervix will be used. For each hrHPV type, chi-square analyses will be used to compare the two HPV vaccination groups with respect to the distribution of that type in the (anus, cervix). Will report the proportion of incident cervical infections that were preceded by anal detection of the same type.
Vaccine-induced antibody titers | Up to week 104
  Will explore the antibody titers for the vaccine type found in the HSIL in these women as compared to those without HSIL caused by that type. Analysis of vaccine titers between those with incident vaccine type HPV infections that persist for 2 or more study visits and those that do not will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, Principal Investigator — University of Witwatersrand, South Africa
Locations (6):
- Moi University School of Medicine, Eldoret, Kenya
- UNC Project Malawi, Lilongwe, Malawi
- South Africa (2):
  - African Cancer Institute at Stellenbosch, Cape Town
  - University of the Witwatersrand, Johannesburg
- Uganda Cancer Institute, Kampala, Uganda
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No